CLINICAL TRIAL: NCT03937648
Title: A Randomized, Double Blind, Placebo-controlled, Single-dose, Dose-escalation Study to Evaluate Pharmacokinetics, Safety, and Tolerability With Oral Administration of Ildong COL-144 Tablet in Korean Healthy Volunteers
Brief Title: Study to Evaluate Pharmacokinetics, Safety, and Tolerability Ildong COL-144 Tablet in Korean Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ID-LAS-101
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- COL-144 50mg (Experimental)
  Interventions: Drug: COL-144 50mg
- COL-144 100mg (Experimental)
  Interventions: Drug: COL-144 100mg
- COL-144 200mg (Experimental)
  Interventions: Drug: COL-144 200mg
- COL-144 400mg (Experimental)
  Interventions: Drug: COL-144 400mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COL-144 50mg — COL-144 50mg
  Arms: COL-144 50mg
Drug: COL-144 100mg — COL-144 100mg
  Arms: COL-144 100mg
Drug: COL-144 200mg — COL-144 200mg
  Arms: COL-144 200mg
Drug: COL-144 400mg — COL-144 400mg
  Arms: COL-144 400mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double blind, Placebo-controlled, Single-dose, Dose-escalation Study to Evaluate Pharmacokinetics, Safety, and Tolerability with Oral Administration of Ildong COL-144 tablet in Korean Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. A healthy adult who is at least 19 years old and less than 50 years old at the time of the screening visit.
2. A person whose body mass index (BMI) is greater than 19 kg/m2 and less than 28 kg/m2 at the time of the screening visit.
3. A person who is medically confirmed to be clinically insignificant in terms of a physical or mental condition by an investigator through a physical examination during the screening period.
4. A person who has agreed to use a combination of effective contraceptive methods or medically appropriate contraceptive methods from the date of administration of the investigational product to the end of the clinical trial (date of test for final safety assessment).
5. A male or female who has agreed not to provide sperm or eggs.
6. A woman whose serum/urine human chorionic gonadotropin (hCG) test results were negative and who is not pregnant or breastfeeding.
7. A person who has voluntarily decided and provided written consent to participate in clinical trials and follow precautions for test subjects.
8. A person who can collect blood and urine during the clinical trial, including follow-up visits.

Exclusion Criteria:

1. A person with a history of gastrointestinal disorders (ex. Crohn's disease, ulcerative colitis, etc.) or surgery (except for simple appendectomy or herniotomy) that may affect the absorption of the investigational product.
2. In addition to Exclusion Criteria 1 above, a person with a history of clinically significant diseases related to allergy, cardiovascular system, peripheral vascular system, skin, mucous membrane, eyes, otolaryngology system, respiratory system, musculoskeletal system, infection, gastrointestinal system, liver, biliary system, endocrine system, kidney, urogenital system, nervous system, psychiatric system, blood, tumor, fracture, and others.
3. A person with genetically caused galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
4. A person with a history of hypersensitivity or clinically significant hypersensitivity to drugs that contain Lasmiditan or ingredients in the same category or other drugs (aspirin and non-steroidal anti-inflammatory drugs, antibiotics, etc.).
5. A person who has a history of drug abuse or whose urine drug screening test result during the screening period came back positive for abusive drug use.
6. A person who has donated partial or full amount of blood within 60 days of the screening visit, who has given blood through apheresis within 30 days, or who has been transfused within 60 days.
7. A person who has been administered with the investigational product or a bioequivalence study drug in another clinical trial or a bioequivalence study within 180 days of the screening visit.
8. A person who has taken a prescription drug, OTC(over the counter drug), herbal medicine, or health-functional food within 14 days of the screening visit.
9. A person who has smoked excessively within 14 days of the screening visit or whose (> 10 cigarettes/day) urine nicotine test result during the screening period came back positive.
10. A person who drank excessively within 14 days of screening visit (> 21 units/week).
11. A person who shows the following results in the vitality sign test during the screening period.

    Systolic blood pressure ≥ 140 (millimeter of mercury) mmHg or <90 mmHg Diastolic blood pressure ≥ 90 mmHg or <60 mmHg Pulse> 100 bpm or < 45 bpm
12. A person who shows the following in the diagnostic test during the screening period.

    * Aspartate aminotransferase (AST) and aminotransferase (ALT) values exceed the upper limit of reference (UNL) by more than 1.5 times.
    * Bilirubin total value exceeds the upper limit of reference (UNL) by more than 1.5 times.
13. A person who tested positive in a blood serum test (hepatitis B test, human immunodeficiency virus (HIV) test, hepatitis C test, syphilis test) during the screening period.
14. A person who showed QTc(Heart rate-corrected QT) > 450 ms or clinically significant abnormalities in a 12-electrode electrocardiogram during the screening period.
15. In addition to Exclusion Criteria 12) to 14), a person who was found to be ineligible to participate in the clinical trials by the diagnostic test or a 12-electrode electrocardiogram.
16. Any other person who is judged to be inadequate to perform the clinical trials by the investigator.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cmax(maximum serum concentration) | 0hours(predose), 0.17hours, 0.33hours, 0.5hours, 0.67hours, 1hours, 1.5hours, 2hours, 2.5hours, 3hours, 4hours, 6hours, 8hours, 12hours, Day2 0hours(24hours), 30hours, Day3 0hours(48hours), 4day 0hours(72hours)
AUClast(rea under the curve from the time of dosing to the last measurable concentration) | 0hours(predose), 0.17hours, 0.33hours, 0.5hours, 0.67hours, 1hours, 1.5hours, 2hours, 2.5hours, 3hours, 4hours, 6hours, 8hours, 12hours, Day2 0hours(24hours), 30hours, Day3 0hours(48hours), 4day 0hours(72hours)
tmax(Time to reach maximum plasma concentration) | 0hours(predose), 0.17hours, 0.33hours, 0.5hours, 0.67hours, 1hours, 1.5hours, 2hours, 2.5hours, 3hours, 4hours, 6hours, 8hours, 12hours, Day2 0hours(24hours), 30hours, Day3 0hours(48hours), 4day 0hours(72hours)
CL/F(Clearance) | 0hours(predose), 0.17hours, 0.33hours, 0.5hours, 0.67hours, 1hours, 1.5hours, 2hours, 2.5hours, 3hours, 4hours, 6hours, 8hours, 12hours, Day2 0hours(24hours), 30hours, Day3 0hours(48hours), 4day 0hours(72hours)